CLINICAL TRIAL: NCT03542656
Title: Application of Amyloid PET in Cerebral Amyloid Angiopathy
Acronym: CAA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201404065MIND
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Cerebral Amyloid Angiopathy; Intracranial Hemorrhages; Alzheimer Disease
Keywords: Stroke; intracerebral hemorrhage; amyoid PET; cerebral amyloid angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Intracranial Hemorrhages; Alzheimer Disease; Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amyloid PET (Experimental): PET/CT
  Interventions: Drug: amyloid PET

INTERVENTIONS:
Drug: amyloid PET — Dynamic PET acquisition for 60 minutes will be acquired after injection of 10 mCi 11C-PiB (39 frames: 8 x 15 seconds, 4 x 60 seconds, 27 x120 seconds).

SUMMARY:
In this project, we will try to enhance the diagnostic potentials of amyloid PET in CAA by combination of dynamic amyloid PET with MRI SWI and MR perfusion images. We will also try to investigate the roles of CAA in patients with drug-related ICH and validate the accuracy of clinical CAA diagnostic criteria. In addition, we will try to study the characteristics of long-term progression of amyloid deposition in CAA patients. This project will enroll 100 patients with ICH, 30 patients with AD, and 30 control subjects. Each patient will receive the above image studies, followed by data analysis and comparison.

DETAILED DESCRIPTION:
Intracranial hemorrhage (ICH) consists of about a quarter of stroke subtype. For elderly, cerebral amyloid angiopathy (CAA) is a common etiology of ICH. In patients with CAA, abnormal beta amyloid protein diffusely deposits at cerebral vasculatures, which disrupts the normal vessel structure and increases the risk of bleeding. The standard diagnosis for CAA requires pathological evidences of amyloid deposition at cerebral arteries. Clinically, a diagnosis of CAA-related ICH is usually only made in an elderly developing cortical or subcortical lobar ICH without undergoing biopsy. Brain images using the SWI sequence of MRI study may show several lobar microbleeds in patients with CAA. However, there is still no direct and precise non-invasive diagnostic tool for CAA until now.

Amyloid PET, using 11C-PiB to image amyloid burden, has been used for detecting the cerebral amyloid protein deposition in patients with Alzheimer's dementia (AD) for years. Recently, amyloid PET has also been applied in diagnosis of CAA. CAA patients showed diffusely increased global PiB retention as compared to control subjects and the distribution of PiB retention is also different from that seen in patients with AD in general. Nevertheless, the applications of amyloid PET in CAA diagnosis are still not well established and many important issues still need to be extensively addressed. For example, amyloid PET sometimes is not able to exactly distinguish CAA patients from control and AD subjects. The roles of CAA in patients with drug-related ICH are still unclear. The accuracy of CAA diagnosis using clinical criteria still needs further validation. In addition, the characteristics for long-term progression of amyloid deposition are still unknown in CAA patients.

In this project, we will try to enhance the diagnostic potentials of amyloid PET in CAA by combination of dynamic amyloid PET with MRI SWI and MR perfusion images. We will also try to investigate the roles of CAA in patients with drug-related ICH and validate the accuracy of clinical CAA diagnostic criteria. In addition, we will try to study the characteristics of long-term progression of amyloid deposition in CAA patients. This project will enroll 100 patients with ICH, 30 patients with AD, and 30 control subjects. Each patient will receive the above image studies, followed by data analysis and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age：above 20 years old with ICH or AD, or control subjects.
* Patient agrees to participate in the study and receive cerebral amyloid PET and MRI SWI and perfusion studies.

Exclusion Criteria:

* Patients could not receive the PET and MRI studies, including but not limited to poor cooperative agitation impeding adequate study, allergy to contrast medium, hemodynamic instability, implantation of cardiac pacemaker, past history of receiving aneurysm clipping, panic mood to MRI study.
* Patients with pregnancy or recently having a plan for pregnancy.
* Patient or family who does not agree to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
PET imaging | in 3 days
  PET data will reconstruct with ordered set expectation maximization, corrected for attenuation, and each frame will be evaluated to verify adequate count statistics and absence of head motion.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No